CLINICAL TRIAL: NCT04109924
Title: A Phase II Study of TAS-102, Irinotecan and Bevacizumab in Pre-Treated Metastatic Colorectal Cancer (TABAsCO)
Brief Title: TAS-102, Irinotecan, and Bevacizumab for the Treatment of Pre-treated Metastatic or Unresectable Colorectal Cancer, the TABAsCO Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Comprehensive Cancer Network (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I 444019
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Results first posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Advanced Colorectal Carcinoma; Metastatic Colon Adenocarcinoma; Metastatic Rectal Adenocarcinoma; Recurrent Colon Adenocarcinoma; Recurrent Colorectal Adenocarcinoma; Recurrent Rectal Adenocarcinoma; Stage III Colon Cancer AJCC v8; Stage III Colorectal Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Colon Cancer AJCC v8; Stage IIIA Colorectal Cancer AJCC v8; Stage IIIB Colorectal Cancer AJCC v8; Stage IIIB Rectal Cancer AJCC v8; Stage IIIC Colon Cancer AJCC v8; Stage IIIC Colorectal Cancer AJCC v8; Stage IV Colon Cancer AJCC v8; Stage IVA Colorectal Cancer AJCC v8; Stage IVA Rectal Cancer AJCC v8; Stage IVB Colon Cancer AJCC v8; Stage IVB Colorectal Cancer AJCC v8; Stage IVB Rectal Cancer AJCC v8; Stage IVC Colon Cancer AJCC v8; Stage IVC Colorectal Cancer AJCC v8; Stage IVC Rectal Cancer AJCC v8; Unresectable Colon Adenocarcinoma; Unresectable Colorectal Carcinoma; Unresectable Rectal Adenocarcinoma
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms; Colorectal Neoplasms | interventions — Irinotecan; Bevacizumab; Disulfides; Trifluridine; trifluridine tipiracil drug combination; Thymidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (irinotecan, bevacizumab, TAS-102) (Experimental): Patients receive irinotecan IV over 90 minutes and bevacizumab IV over 10 minutes on days 1 and 15. Patients also receive trifluridine and tipiracil hydrochloride PO BID on days 2-6 and 16-20. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Irinotecan; Biological: Bevacizumab; Drug: Trifluridine and Tipiracil Hydrochloride

INTERVENTIONS:
Drug: Irinotecan — Given IV
  Other Names: (+)-(4S)-4; 11-diethyl-4-hydroxy-9-[(4-piperidino-piperidino)carbonyloxy]-1H-pyrano[3'',4'':6,7]indolizino[1,2-b]quinol-3,14,(4H,12H)-dione; (+)-7-ethyl-10-hydroxycamptothecine 10-[1,4''-bipiperidine]-1''-carboxylate,; 616348,; 7-ethyl-10-[4-(1-piperidino)-1-piperidino]carbonyloxycamptothecin; 728073; 97682-44-5
Biological: Bevacizumab — Given IV
  Other Names: 216974-75-3; 704865; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain,; Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501
Drug: Trifluridine and Tipiracil Hydrochloride — Given PO
  Other Names: 733030-01-8; Lonsurf; TAS 102; TAS-102; Thymidine; Alpha; Mixt. with 5-Chloro-6-((2-imino-1-pyrrolidinyl)methyl)-2,4(1H,3H)-pyrimidinedione Monohydrochloride; Tipiracil Hydrochloride Mixture with Trifluridine; Trifluridine/Tipiracil,

SUMMARY:
This phase II trial studies how well TAS-102, irinotecan, and bevacizumab work in treating patients with pre-treated colorectal cancer that has spread to other places in the body (metastatic) or cannot be removed by surgery (unresectable). Drugs used in chemotherapy, such as TAS-102, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Irinotecan may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with bevacizumab, may induce changes in body's immune system and may interfere with the ability of tumor cells to grow and spread. Giving TAS-102, irinotecan, and bevacizumab may work better in treating patients with colorectal cancer compared to traditional chemotherapy and bevacizumab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the median progression free survival (PFS) benefit of leucovorin calcium, 5-fluorouracil, and irinotecan (FOLFIRI) naive patients treated with trifluridine and tipiracil hydrochloride (TAS-102) + irinotecan + bevacizumab as compared to historic control groups treated with FOLFIRI + bevacizumab.

SECONDARY OBJECTIVE:

I. Estimate the objective response rate (ORR), median overall survival (OS), and adverse event (AE) profile.

OUTLINE:

Patients receive irinotecan intravenously (IV) over 90 minutes and bevacizumab IV over 30-90 minutes on days 1 and 15. Patients also receive trifluridine and tipiracil hydrochloride orally (PO) twice daily (BID) on days 2-6 and 16-20. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Advanced colorectal cancer (metastatic or unresectable): Histologically or cytological proven adenocarcinoma of the colon or rectum which is metastatic or otherwise incurable
* Prior treatment with a fluoropyrimidine (5-fluorouracil [5-FU] or capecitabine) and oxaliplatin in the metastatic/unresectable setting OR, recurrence within 12 months of adjuvant therapy with a regimen that included oxaliplatin
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Hemoglobin >= 9 g/dL
* Absolute neutrophil count >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Creatinine < 1.5 upper limit of normal (ULN) or if >= 1.5 x ULN creatinine clearance (CRCL) >= 30 mL/min (by Cockcroft-Gault)
* Bilirubin < 1.5 x ULN
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 2.5 x ULN or =< 5 x ULN if with hepatic metastases
* Have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria present
* Participants of child-bearing potential must agree to use adequate contraceptive methods (e.g., hormonal or barrier method of birth control; abstinence) prior to study entry. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately
* Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Prior treatment with TAS-102 or irinotecan
* Anti-cancer therapy within 2 weeks of the planned first dose of study medication
* Unresolved toxicities from prior therapy of > grade 1, excluding alopecia or similar toxicities which are not deemed to be clinically significant or put the participant at greater risk. Grade 2 neuropathy is permitted
* Major surgery within 4 weeks of anticipated start of therapy
* Uncontrolled hypertension: systolic blood pressure >= 150, diastolic blood pressure >= 100
* Unstable angina, symptomatic congestive heart failure or cardiac arrhythmia requiring anti-arrhythmic therapy (beta-blockers, calcium channel blockers and digoxin are allowed)
* Arterial or venous thrombotic or embolic events within 3 months of study initiation, unless well controlled on stable anti-coagulation for >= 2 weeks. This excludes uncomplicated catheter associated venous thrombosis
* History of cerebrovascular or myocardial ischemia within 6 months of initiation
* National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0 grade 3 or greater hemorrhage within the past 4 weeks
* Proteinuria >= 2+, unless 24 hour urine collection demonstrates =< 1 g of protein OR spot protein: creatinine demonstrates a ratio of =< 1
* Untreated brain metastases
* History of abnormal glucuronidation of bilirubin (Gilbert's syndrome)
* History of second primary malignancy within 3 years prior to enrollment, excluding in-situ cervical carcinoma, non-melanoma skin cancer or malignancy of equivalent risk which is highly unlikely to require systemic treatment in the next 2 years
* Have known active infection which would heighten the risk of complications
* Pregnant or nursing female participants
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-12-27 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Fountzilas, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Boland PM, Mukherjee S, Imanirad I, Vijayvergia N, Cohen SD, Gupta M, Iyer RV, Bakin A, Wang J, Chatley S, Cahill B, Vadehra D, Attwood K, Hochster HS, Fountzilas C. TAS-102, Irinotecan, and bevacizumab in pre-treated metastatic colorectal cancer (TABAsCO), a phase II clinical trial. Br J Cancer. 2024 Nov;131(8):1290-1297. doi: 10.1038/s41416-024-02845-x. Epub 2024 Sep 7. PMID 39244627

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Irinotecan, Bevacizumab, TAS-102)
Started | 42
Completed | 35
Not Completed | 7
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — Incomplete baseline imaging | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Irinotecan, Bevacizumab, TAS-102)
Number analyzed (Participants) | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 26
  >=65 years | 16
Age, Continuous [Median (Full Range); unit: years] | 59 [40.2 to 85.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 32
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS)
Description: Will be assessed via the Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 guidelines. The PFS will be summarized using standard Kaplan-Meier methods, where estimates of the median PFS and 6/12-month PFS rates will be obtained with 90% confidence intervals.
Time Frame: Medical record review will be performed approximately every 6 months, for up to 2 years, post treatment up to 4 years
Population: Only 35 patients completed treatment. The primary outcome(i.e. Median progression free survival (PFS)) analysis is based on these 35 patients who completed treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Irinotecan, Bevacizumab, TAS-102)
Number analyzed (Participants) | 35
months | 7.9 [5.6 to 11.4]

2. Secondary Outcome: Number of Participants With Complete Response, Partial Response, Stable Disease and Progressive Disease
Description: Patients receive irinotecan IV over 90 minutes and bevacizumab IV over 10 minutes on days 1 and 15. Patients also receive trifluridine and tipiracil hydrochloride PO BID on days 2-6 and 16-20. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Irinotecan: Given IV
  Bevacizumab: Given IV
  Trifluridine and Tipiracil Hydrochloride: Given PO
Time Frame: Medical record review will be performed approximately every 6 months, for up to 2 years, post treatment up to 4 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Irinotecan, Bevacizumab, TAS-102)
Number analyzed (Participants) | 35
Participants
  CR | 1
  PR | 6
  SD | 20
  PD | 8

3. Secondary Outcome: Median Overall Survival (OS)
Description: OS will be summarized using standard Kaplan-Meier methods; where estimates of the median survival are obtained with 90% confidence intervals
Time Frame: Medical record review will be performed approximately every 6 months, for up to 2 years, post treatment up to 4 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Irinotecan, Bevacizumab, TAS-102)
Number analyzed (Participants) | 35
months | 16.7 [11.8 to 22.8]

4. Secondary Outcome: Disease-specific Survival (DSS)
Description: DSS will be summarized using standard Kaplan-Meier methods; where estimates of the median survival and 12-month rates are obtained with 90% confidence intervals.
Time Frame: Medical record review will be performed approximately every 6 months, for up to 2 years, post treatment up to 4 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (Irinotecan, Bevacizumab, TAS-102)
Number analyzed (Participants) | 35
months | 16.7 [11.8 to 22.8]

5. Secondary Outcome: Aggregate Rates of Adverse Events
Description: measured by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 and recorded to objectively measure toxicities of the combination therapy. Treatment related adverse events (as per CTCAE v5.0) will be summarized by grade using frequencies and relative frequencies. Only grade 4 and 5 adverse events are reported here.
Time Frame: Follow-up safety evaluations will occur 30 days (± 3 days) after last dose of study drug or until resolution of any drug related toxicity (telephone contact is acceptable), through study completion , an average of 3.5 years work
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Irinotecan, Bevacizumab, TAS-102)
Number analyzed (Participants) | 42
Participants
  developed grade 4/5 adverse events | 9
  Not developed 4/5 adverse events | 33

ADVERSE EVENTS:
Time Frame: Follow-up safety evaluations will occur 30 days (± 3 days) after last dose of study drug or until resolution of any drug related toxicity (telephone contact is acceptable), through study completion, an average of 3.5 years, up to 4 years
Description: An adverse event or adverse experience (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Therefore, an AE can be ANY unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not considered related to the medicinal (investigational) product
Arm/Group | Treatment (Irinotecan, Bevacizumab, TAS-102)
All-Cause Mortality (participants affected / at risk) | 33/42
Serious Adverse Events (participants affected / at risk) | 12/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Irinotecan, Bevacizumab, TAS-102) (N=42)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Colitis (Gastrointestinal disorders) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Endocarditis infective (Infections and infestations) | 1 (1)
Pelvic infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Headache (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Irinotecan, Bevacizumab, TAS-102) (N=42)
Anemia (Blood and lymphatic system disorders) | 14 (14)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Anal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (7)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 30 (30)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 28 (28)
Proctitis (Gastrointestinal disorders) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (14)
Fatigue (General disorders) | 26 (26)
Pain (General disorders) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Shingles (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 7 (7)
Intestinal stoma site bleeding (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 6 (6)
Neutrophil count decreased (Investigations) | 32 (32)
Platelet count decreased (Investigations) | 10 (10)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 11 (11)
Anorexia (Metabolism and nutrition disorders) | 14 (14)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (15)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2)
Hot flashes (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT04109924/Prot_SAP_000.pdf